CLINICAL TRIAL: NCT00364429
Title: Investigation of the NMDA Receptor System in Man as a Potential Surrogate Marker for Deficit Syndrome in Schizophrenia: a [123]I-CNS 1261 Single Photon Emission Tomography (SPET) Study
Brief Title: SPECT Investigation Of The NMDA Receptor System In Healthy Volunteers And Patients With Schizophrenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: terminated
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 102747
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia
Keywords: schizophrenic patients; SPET; NMDA receptor; ligand [123]I-CNS 1261
MeSH Terms: conditions — Schizophrenia | interventions — Lorazepam; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: [123]I-CNS 1261 — Study Drug
Drug: Lorazepam — Study Drug
Drug: Risperidone — Study Drug
  Other Names: [123]I-CNS 1261; Lorazepam

SUMMARY:
This study was designed to compare the [123]I-CNS 1261 binding to NMDA receptor between healthy volunteers and different subgroups of schizophrenic patients. Investigation of the potential influence of antipsychotic and concomitant medication on [123I] CNS 1261 binding is also relevant.Fifteen healthy subjects (male and female of non-child bearing potential) will be recruited and 40 schizophrenic patients divided in 3 subgroups as indicated before: Subgroup a) treatment-naive, (n=10); Subgroup b) on stable treatment with risperidone (without criteria of deficit syndrome on the SDS scale, (n=15);Subgroup c) on stable treatment with risperidone fitting criteria of deficit syndrome on the SDS scale, (n=15).

ELIGIBILITY:
Inclusion criteria:

* Right-handed
* Smoker
* Healthy volunteer or schizophrenic patients as diagnosed by DSM IV criteria.
* Treatment naive patients or with Risperidone treatment for 2 months that have not received any depot neuroleptic during the last year.
* Women of childbearing potential must agree to acceptable method of birth control.

Exclusion criteria:

* Any clinically or laboratory significant abnormality.
* Subjects receiving a radiation dose from other activities of more than 10 mSv over any 3 year period.
* Heart pacemaker, metallic prosthesis or other metallic body implants.
* History or presence of CNS conditions.
* History of substance dependence.
* History of or suffers from claustrophobia.
* Positive test for HBV (hepatitis B virus), HCV (hepatitis C virus) or HIV.
* Pregnant or lactating women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2005-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
CNS (Central Nervous System) 1261 binding differences in healthy volunteers and 3 different predefined subgroups of schizophrenic patients and in the 3 different subgroups of schizophrenic patients. | throughout the study

SECONDARY OUTCOMES:
Effect of treatment with risperidone and lorazepam in inducing changes on [123]I CNS 1261 binding, and its relationship with the plasma concentration of administered drugs and with Psychopathological scales scores. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Barcelona, Spain